CLINICAL TRIAL: NCT00520091
Title: A Pilot Study of the Biologic Efficacy and Safety of the Addition of Celecoxib to a Program of Induction Chemotherapy and Neo-Adjuvant Chemo-Radiotherapy for the Treatment of Esophageal Cancer
Brief Title: Irinotecan, Cisplatin, and Radiation Therapy With or Without Celecoxib in Treating Patients With Stage II, Stage III, or Stage IV Esophageal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 0203; CDR0000561610 (Other: NCI PDQ identifier); NCT00280124 (obsolete NCT alias)
Record Dates: First submitted 2007-08-21; First posted 2007-08-23 (Estimated); Last update posted 2012-05-18 (Estimated); Status verified 2012-05

CONDITIONS: Esophageal Cancer
Keywords: adenocarcinoma of the esophagus; squamous cell carcinoma of the esophagus; stage II esophageal cancer; stage III esophageal cancer; stage IV esophageal cancer
MeSH Terms: conditions — Esophageal Neoplasms; Adenocarcinoma Of Esophagus; Esophageal Squamous Cell Carcinoma | interventions — Irinotecan; Cisplatin; Celecoxib; Radiation; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort 1 (Active Comparator): Induction chemotherapy and chemoradiation without celecoxib
  Interventions: Drug: CPT- 11; Drug: Cisplatin; Radiation: Radiation; Procedure: Surgery
- Cohort 2 (Experimental): Induction chemotherapy and chemoradiation with celecoxib
  Interventions: Drug: CPT- 11; Drug: Cisplatin; Drug: Celecoxib; Radiation: Radiation; Procedure: Surgery

INTERVENTIONS:
Drug: CPT- 11 — 65mg/m2 given on days 1, 8 ,22 and 29 prior to surgery
  Other Names: Irinotecan
Drug: Cisplatin — Cisplatin 30mg/m2 will be administered on days 1, 8, 22 and 29 prior to surgery
  Other Names: Cis-diammine-dichloro-platinum
Drug: Celecoxib — 400 mg, orally, twice per day beginning on day minus 3 and continue until the end of chemoradiation with CPT-11 and Cisplatin
  Arms: Cohort 2
Radiation: Radiation — 4,500 cGy in 180 cGy fractions 5 days per week, over a period of 5 weeks
Procedure: Surgery — Surgery will occur prior to chemoradiation therapy for those patients with resectable disease

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as irinotecan and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Celecoxib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving chemotherapy and radiation therapy together with celecoxib may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving irinotecan and cisplatin together with radiation therapy with or without celecoxib works in treating patients with stage II, stage III, or stage IV esophageal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To measure the rates of cellular apoptosis and proliferation at baseline and during chemoradiotherapy with and without celecoxib using biopsy samples from patients with stage II, III, or IV esophageal cancer.
* To determine if an acceptable rate of pathologic complete remission can be achieved in a subset of patients with potentially resectable esophageal cancer.

Secondary

* To assess the safety of the addition of daily celecoxib to chemoradiotherapy.
* To estimate the median overall survival in a subset of patients with resectable disease.
* To quantitate expression of cyclooxygenase (COX)-2 and formation of prostaglandin E2 (PGE2) in patients with esophageal cancer.
* To assess the ability of celecoxib to decrease formation of PGE2 in tumor tissue by measuring pre- and post-treatment tumor concentrations of PGE2.
* To quantitate downstream effects of inhibition of COX-2 function in the setting of treatment with chemotherapy.
* To measure the radiographic response rate in patients with unresectable esophageal cancer.

OUTLINE: This is a multicenter study. Patients are sequentially enrolled into 1 of 2 treatment groups.

* Group 1: Patients receive cisplatin IV over 1 hour and irinotecan hydrochloride IV over 90 minutes on days 1, 8, 22, 29, 43, 50, 64, and 71. Patients also undergo radiotherapy once daily 5 days a week for 5 weeks beginning on day 43.
* Group 2: Patients receive chemoradiotherapy as in group 1. Patients also receive oral celecoxib twice daily beginning 3 days before the initiation of chemotherapy and continuing until the completion of chemoradiotherapy.

In both groups, patients with potentially resectable disease undergo surgery no more than 12 weeks after completion of chemoradiotherapy.

Endoscopic tumor biopsy specimens are collected at baseline and on day 3 of radiotherapy. Samples are analyzed for cyclooxygenase (COX)-2 gene and protein expression; PGE2 secretion; apoptotic activity; caspase-3 activation; cytochrome c translocation; VEGF mRNA quantitation; and cellular proliferation. Laboratory techniques used include RT-PCR, IHC, enzyme immunoassay, TUNEL assay, colorimetric assay, and northern blotting.

After completion of study treatment, patients are followed every 3 months for 2 years, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 34 patients (8-10 in group 1 and 24 in group 2) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Biopsy proven squamous cell carcinoma or adenocarcinoma of the esophagus

  * Lesions including the gastroesophageal junction allowed provided the tumor involves less than 2 cm of gastric cardia
* Meets 1 of the following criteria:

  * Clinical stage II, III, or IV disease AND planning to receive chemoradiotherapy either for preoperative or palliative indications (group 1)

    * Suitable candidate for bimodality (palliative intent) or trimodality (curative intent) therapy
  * Clinical stage II or III disease AND candidate to receive chemoradiotherapy for preoperative indication followed by planned esophagectomy or esophagogastrectomy (group 2)

    * Suitable candidate for trimodality (curative intent) therapy
* No tracheoesophageal fistula on bronchoscopy

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy > 3 months (group 1)
* Not pregnant
* Adequate nutrition
* WBC ≥ 4,000/μL
* ANC ≥ 1,500/μL
* Platelet count ≥ 100,000/μL
* Serum creatinine ≤ 1.5 mg/dL
* Bilirubin ≤ 1.5 mg/dL
* No other prior or concurrent malignancy other than curatively treated carcinoma in situ of the cervix; localized prostate cancer that was previously treated with local therapy more than 2 years ago with a PSA of less than 4 ng/mL; basal cell carcinoma of the skin; or superficial transitional cell carcinoma of the bladder

  * Patients who have had a prior malignancy are eligible if they have been free of disease for ≥ 5 years
* No serious medical or psychiatric illnesses that would preclude giving informed consent or otherwise limit survival to less than 2 years
* No history of known NSAID-induced gastrointestinal bleeding
* No current peptic ulcer disease
* No active coronary artery disease
* No myocardial infarction or cerebrovascular accident within the past 3 months
* No history of refractory congestive heart failure or cardiomyopathy

PRIOR CONCURRENT THERAPY:

* More than 1 week since prior major surgery (group 1)
* More than 2 weeks since prior major surgery (group 2)
* No prior chemotherapy or radiotherapy
* More than 30 days since prior cyclooxygenase-2 inhibitors (selective or non-selective), including, but not limited to, any of the following:

  * Acetylsalicylic acid (aspirin)
  * Piroxicam
  * Diclofenac
  * Meloxicam
  * Indomethacin
  * Fenoprofen
  * Sulindac
  * Flurbiprofen
  * Tolmetin
  * Ibuprofen
  * Celecoxib
  * Ketoprofen
  * Rofecoxib
  * Ketoprofen ER
  * Valdecoxib
  * Naproxen
  * Meclofenamate
  * Oxaprozin
  * Mefenamic acid
  * Etodolac
  * Nabumetone
  * Ketorolac
* No concurrent seizure medications
* No concurrent amifostine or other such agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2005-03; Primary Completion 2006-11 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Rates of cellular apoptosis and proliferation | 5 weeks
  Measure the rates of cellular apoptotis and proliferation in esophageal cancers from biopsy samples pre-study and during chemoradiation with and without celecoxib therapy
Rate of pathologic complete remission in patients with resectable disease | 4 years
  To determine if an acceptable rate of pathologic complete remissions can be achieved in a cohort of patients with potentially resectable esophageal carcinoma

SECONDARY OUTCOMES:
Number of subjects experiencing adverse events | 30 days post radiation
  Adverse events/toxicity will graded per the CTCAE criteria
Median overall survival of patients with resectable disease | 4 years
  Follow up for survival will occur at 3 month intervals during the first two years, then every 6 months during years 3 and 4.
Formation of prostaglandin E2 (PGE2) in tumor tissue | 12 weeks
  The ability of celecoxib to decrease formation of prostaglandin E2 (PGE2) in tumor tissue will be analyzed using a Wilcoxon signed rank test on the difference (log scale) of the pre- and post-treatment tumor concentrations of PGE2
Downstream effects of inhibition of cyclooxygenase 2 function | 12 weeks
  A difference in location of the mRNA expression of the two cohorts will be tested for using the Wilcoxon rank sum test. A difference in the immunohistochemistry staining of the two cohorts will be tested for using polytomous logistic regression
Response Rate | 4 years
  Radiographic repsonse will be measured using RECIST critera in patients with unresectable esophageal cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Bert H. O'Neil, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center